CLINICAL TRIAL: NCT05860465
Title: A Phase II/III Study of SPH4336 in Combination With Endocrine Therapy in the Treatment of HR-positive, HER2-negative Locally Advanced or Metastatic Breast Cancer That Progressed on CDK4/6 Inhibitor Combined With Endocrine Therapy
Brief Title: Safety and Efficacy of SPH4336 in Combination With Endocrine Therapy in the Treatment of Locally Advanced or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH4336-302
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPH4336 Tablets (Experimental): SPH4336 Tablets; Letrozole tablets; Fulvestrant injection
  Interventions: Drug: SPH4336 Tablets
- SPH4336 Tablets Placebo (Placebo Comparator): SPH4336 Tablets Placebo; Letrozole tablets; Fulvestrant injection
  Interventions: Drug: SPH4336 Tablets Placebo

INTERVENTIONS:
Drug: SPH4336 Tablets — SPH4336 Tablets ：Administered by oral; Letrozole tablets：Administered by oral; Fulvestrant injection：Administered by intravenous infusion
  Arms: SPH4336 Tablets
Drug: SPH4336 Tablets Placebo — SPH4336 Tablets Placebo ：Administered by oral; Letrozole tablets：Administered by oral; Fulvestrant injection：Administered by intravenous infusion
  Arms: SPH4336 Tablets Placebo

SUMMARY:
This study evaluated the safety and efficacy of SPH4336 in combination with endocrine therapy in the treatment of locally advanced or metastatic breast cancer that progressed on CDK4/6 inhibitor combined with endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate in this study, completely understand this study, and voluntarily sign the informed consent form (ICF).
2. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 or 1.
3. Life expectancy ≥ 3 months.
4. Patients with locally advanced or metastatic breast cancer who are unable to receive radical surgeries/other local therapies.
5. At least one measurable lesion.
6. Laboratory test results meet the relevant requirements for organ function.
7. Subjects who agree to take effective contraceptive measures.

Exclusion Criteria:

1. Inflammatory breast cancer.
2. Patients unsuitable for endocrine therapy at the investigator's discretion.
3. History of other malignancies prior to the start of study treatment.
4. Patients with known metastases to central nervous system.
5. Taking anti-tumor traditional Chinese patent medicines at the time of signing the ICF.
6. Patients who underwent a surgery prior to the start of study treatment, and have not yet recovered from adverse reactions of the surgery.
7. Patients who participated in a clinical trial and received other investigational drugs before the start of study treatment.
8. Pregnant or lactating women.
9. History of myocardial infarction, unstable angina pectoris, severe arrhythmia, and symptomatic congestive heart failure before the start of study treatment; ≥ NYHA (New York Heart Association) Class II; mean QTc interval ≥ 470 ms before the start of study treatment; left ventricular ejection fraction ≤ 50% before the start of study treatment.
10. History of ischemic stroke or severe thromboembolic disease before the start of study treatment.
11. Hepatitis B surface antigen positive and HBV (Hepatitis B Virus) DNA > 2,000 IU/mL or > 104 copies/mL; HCV (Hepatitis C Virus) antibody positive and HCV RNA positive; or known HIV infection.
12. History of severe allergic diseases, history of severe drug allergies, or known allergy to any ingredient of the investigational product.
13. Presence of diseases or conditions that may impact drug administration or gastrointestinal absorption before the start of study treatment.
14. Presence of uncontrolled infections before the start of study treatment.
15. Known history of drug abuse, excessive drinking, or illegal drug use; history of confirmed neurological or mental disorders.
16. Presence of other diseases that the risks of receiving the study treatment outweigh its benefits, as determined by the investigator, or any other reason for which patients are ineligible for the study as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 254 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Approximately 3years
  tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.
Progression-free survival (PFS) | Approximately 3years
  from the start date of study treatment to the date of progression disease or death , whichever occurred first.

SECONDARY OUTCOMES:
Cmax | Approximately 3years
  PK (Pharmacokinetics) parameters
Tmax | Approximately 3years
  PK (Pharmacokinetics) parameters
Disease control rate (DCR) | Approximately 3years
  DCR was defined as the percentage of patients who have achieved complete response, partial response and stable disease
Duration of remission (DOR) | Approximately 3years
  DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response to the date of disease progression per RECIST v1.1 or death from any cause
Overall Survival (OS) | Approximately 8years
  Determination of the overall survival times of all patients
Safety and tolerability of the combination therapy since the start of any study treatment. | Approximately 3years
  Adverse event type, incidence, duration, correlation with study drug

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Affiliated Cancer Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Liuzhou people's Hospital, Liuchow, Guangxi
  - Anyang Cancer Hospital, Anyang, He'nan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, He'nan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University cancer Hospital, Harbin, Heilongjiang
  - Xiangyang Cancer Hospital, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - The second people's hospital of neijiang, Neijiang, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang cancer Hospital, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Fujian Cancer Hospital, Fuzhou
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - Shenzhen Hospital of University of Hong Kong, Shenzhen
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin